CLINICAL TRIAL: NCT05217537
Title: A Phase 1, Open-Label, Multi-Center Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Intravenous and Oral Doses of Omadacycline in Pediatric Subjects With Suspected or Confirmed Bacterial Infections
Brief Title: Study to Evaluate the PK of IV and PO Omadacycline in Children and Adolescents With Suspected or Confirmed Bacterial Infections
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Paratek Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PTK0796-PEDPK-20110
Record Dates: First submitted 2021-12-15; First posted 2022-02-01 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — omadacycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (adolescents) (Experimental): 12 to < 18 years of age
  Interventions: Drug: Omadacycline Injection [Nuzyra]; Drug: Omadacycline Oral Tablet
- Cohort 2 (children) (Experimental): 8 to < 12 years of age
  Interventions: Drug: Omadacycline Injection [Nuzyra]; Drug: Omadacycline Oral Tablet

INTERVENTIONS:
Drug: Omadacycline Injection [Nuzyra] — Single dose of 100 mg omadacycline IV in 100 mL of normal saline
  Other Names: NUZYRA
Drug: Omadacycline Oral Tablet — Single dose of 300 mg omadacycline PO (2 x 150 mg tablets)
  Other Names: NUZYRA

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of a single dose of intravenous or oral omadacycline in children and adolescents with suspected or confirmed bacterial infections.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, age 8 to < 18 (inclusive) who have written and signed parental/legal authorized representative (LAR) informed consent and pediatric assent.
* Currently hospitalized with a suspected or confirmed bacterial infection and receiving or planned to receive systemic antibiotic therapy other than omadacycline.
* Weight within the 5th and 95th percentile for age and sex.
* Subjects must not be pregnant or nursing at the time of enrollment, and must agree to use a highly effective birth control method during the study

Exclusion Criteria:

* Evidence of a medical condition that may pose a safety risk or impair study participation.
* Confirmed or suspected SARS-CoV-2 infection.
* Has a history of hypersensitivity or allergic reaction to any tetracycline antibiotic.
* Has received an investigational drug within the past 30 days.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Characterize the PK of a single IV dose of omadacycline in children and adolescents 8 to < 18 years of age with suspected or confirmed bacterial infections | Pre-dose, and 0.5, 1, 2, 8, and 24 hours post-dose
  Plasma concentrations of omadacycline for PK analysis from Day 1 to Day 2
Characterize the PK of a single PO dose of omadacycline in children and adolescents 8 to < 18 years of age with suspected or confirmed bacterial infections | Pre-dose, and 1, 2, 3, 8, and 24 hours post-dose
  Plasma concentrations of omadacycline for PK analysis from Day 1 to Day 2

SECONDARY OUTCOMES:
Adverse events and serious adverse events | From the time of signing the informed consent form up to study completion visit (up to 9 days)
  Incidence, severity, and type of adverse events and serious adverse events
Clinical laboratory tests | From the time of signing the informed consent form up to study completion visit (up to 9 days)
  Number of participants with abnormal clinical laboratory tests
Vital signs | From the time of signing the informed consent form up to study completion visit (up to 9 days)
  Number of participants with clinically significant changes from baseline in vital signs
Physical examination | From the time of signing the informed consent form up to study completion visit (up to 9 days)
  Number of participants with clinically significant abnormal physical examination findings

CONTACTS AND LOCATIONS:
Overall Officials: Amy Manley, Study Director — Paratek Pharmaceuticals Inc
Locations (9):
- United States (9):
  - Site 109, Little Rock, Arkansas
  - Site 112, Long Beach, California
  - Site 107, Orange, California
  - Site 114, Aurora, Colorado
  - Site 105, Chicago, Illinois
  - Site 111, Greenville, North Carolina
  - Site 106, Cleveland, Ohio
  - Site 113, Philadelphia, Pennsylvania
  - Site 108, Houston, Texas

IPD SHARING:
Plan to Share IPD: No